CLINICAL TRIAL: NCT05203406
Title: The Cardio-Sarcopenia Study
Status: Active, not recruiting | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/2263
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Ageing; Physical Activity; Older Adults; Sarcopenia
Keywords: aging; cardiovascular; skeletal muscle; sarcopenia; prevention; digital technology
MeSH Terms: conditions — Motor Activity; Sarcopenia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The use of surrogate markers such as body mass index (BMI) as a target outcome of physical activity may not be appropriate in older adults who are at risk of muscle sarcopenia. In the presence of sarcopenia, reductions in body weight may lead to lower BMI values. We have previously found deleterious changes in cardiac structure and function among sarcopenic older adults, raising a possible biological syndrome of 'cardio-sarcopenia'. In this study, we will investigate the impact of physical activity on temporal changes in cardiac and skeletal muscle , and BMI, over six- to twelve month period, on older adults with this syndrome. By targeting the cardio-sarcopenic phenotype as a modifiable risk factor that may be altered by physical activity, the results will provide new knowledge into retarding deleterious consequences of cardiovascular ageing. This new target challenges the paradigm of using BMI as an anthropometric marker in health prevention. If proven, this will dramatically change primary prevention targets among older adults, justifying the use of cardio-sarcopenia as a rational anthropometric target.

DETAILED DESCRIPTION:
This study builds upon our group's work where we characterized cardiovascular and skeletal muscle structure and function of community-based older adults. In this proposal, we will identify n=100 participants with cardio-sarcopenia phenotype. Comparing between participants with baseline low versus high levels of physical activity, we will investigate temporal changes in their cardiovascular, skeletal muscle, biomarkers and BMI data, over a six- to twelve month period. Physical activity will include subjective self-reported physical activities and objective measures of aerobic capacity. Their physical activity levels will be verified bi-monthly via physical activity and cardiac health application that measures these markers. Pertinent fluctuations in diet, lifestyle, risk factors and biomarkers will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* >=21 years of age

Exclusion Criteria:

* Unable to provide written informed consent to participate in the study.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are recruited through population based studies (SingHealth IRB 2018/3173) who have agreed to be contacted for future studies.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2051-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in cardio-sarcopenia | Six to twelve months
  To compare differences in skeletal muscle (structure and function) and CV imaging markers, between older adults with low versus high physical activity levels, over time, at baseline and at six- to twelve months

SECONDARY OUTCOMES:
Changes in body mass index (BMI) | Six to Twelve months
  To study rates of changes in body mass index in relation to changes in cardio-sarcopenia.

OTHER OUTCOMES:
Changes in cardiac function as assessed by personalized digital health application. | Six to Twelve month
  To test feasibility and utility of using cardiac health application to input markers of physical activity, deriving automated feedback about cardiac function.

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keng BMH, Gao F, Teo LLY, Lim WS, Tan RS, Ruan W, Ewe SH, Koh WP, Koh AS. Associations between Skeletal Muscle and Myocardium in Aging: A Syndrome of "Cardio-Sarcopenia"? J Am Geriatr Soc. 2019 Dec;67(12):2568-2573. doi: 10.1111/jgs.16132. Epub 2019 Aug 16. PMID 31418823